CLINICAL TRIAL: NCT02879227
Title: Phase II of Radiochemotherapy in Elderly Patients With Oesophagus Cancer
Brief Title: Radiochemotherapy in Elderly Patients With Oesophagus Cancer
Acronym: Chronos
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P/2009/79
Record Dates: First submitted 2016-08-03; First posted 2016-08-25 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Esophagus Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Cisplatin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm Cisplatin (Active Comparator): Radiotherapy 50 Gy with cisplatin 75 mg/2 Day 1 and day 22 (2)
  Interventions: Drug: Cisplatin
- Arm Oxaliplatin (Experimental): Radiotherapy 50Gy Oxaliplatin 85mg/m2 every 2 weeks, (6)
  Interventions: Drug: Oxaliplatin

INTERVENTIONS:
Drug: Cisplatin — Arm cisplatin : 75mg/m2, day n*1 and day n*22, And radiotherapy 50 Gy, 2Gy/f
  Other Names: Arm Cisplatin
  Arms: Arm Cisplatin
Drug: Oxaliplatin — 85 mg/m2 every 2 weeks, 6 times And radiotherapy 50 Gy, 2Gy/f
  Other Names: Arm Oxaliplatin
  Arms: Arm Oxaliplatin

SUMMARY:
Phase II study of radiochemotherapy for elderly patients with oesophagus cancer.

DETAILED DESCRIPTION:
Phase II study of radiochemotherapy for elderly patients with oesophagus cancer with Radiotherapy = 50 Gy, 2Gy/f ans chemotherapy with 2 arms arm Cisplatin = Cisplatin 75mg/m2 J1J22 or arm Oxaliplatine = oxaliplatine 85mg/m2 every 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 75 or more with oesophagus cancer (squamous or adenocarcinoma), fit to treat

Exclusion Criteria:

* previous radiotherapy
* no fit to treat

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Feasibility of treatment: Number of patients with completed treatment | 6 weeks after end of the radiochemotherapy
  number of patient with completed treatment

SECONDARY OUTCOMES:
Tumoral response | 6 weeks after end of the radiochemotherapy
  tumoral evaluation at 6 weeks after the treatment
Quality of life | 6 weeks after end of the radiochemotherapy
  QLQC30
Quality of life | 6 weeks after end of the radiochemotherapy
  ELD14

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Servagi-Vernat S, Bosset M, Crehange G, Buffet-Miny J, Puyraveau M, Maingon P, Mercier M, Bosset JF. Feasibility of chemoradiotherapy for oesophageal cancer in elderly patients aged >or=75 years: a prospective, single-arm phase II study. Drugs Aging. 2009;26(3):255-62. doi: 10.2165/00002512-200926030-00006. PMID 19358620
- [Result] Servagi-Vernat S, Crehange G, Roullet B, Guimas V, Maingon P, Puyraveau M, Bosset JF. Phase II Study of a Platinum-Based Adapted Chemotherapy Regimen Combined with Radiotherapy in Patients 75 Years and Older with Esophageal Cancer. Drugs Aging. 2015 Jun;32(6):487-93. doi: 10.1007/s40266-015-0275-8. PMID 26038198